CLINICAL TRIAL: NCT00200382
Title: Phase II Study to Evaluate the Efficacy and Safety of Therapy With PS 341 in Patients With Advanced Stage Non Small Cell Lung Cancer
Brief Title: Phase II Study of Therapy With PS 341 in Patients With Advanced Stage Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study did not achieve the statistical success to continue.
Sponsor: Rasim Gucalp (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Rasim Gucalp, Prof. Dept of Medicine (Oncology), Montefiore Medical Center
Organization: Montefiore Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-05-123
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bortezomib

INTERVENTIONS:
Drug: PS-341 (Velcade-drug)

SUMMARY:
The purpose of this study is to develop new treatments that will hopefully result in the relief of symptoms and prolongation of life. For this reason, your doctors have offered you treatment with a new experimental drug called PS 341.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have confirmed NSCLC (squamous, adeno- and large cell anaplastic carcinoma)stage III B or Stage IV.

No prior chemotherapy regimen Patients must have adequate organ and marrow function

Exclusion Criteria:

* Untreated symptomatic brain metastasis Patients with known HIV positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2004-05 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Response rate

CONTACTS AND LOCATIONS:
Overall Officials: Rasim Gucalp, M.D., Study Chair — Montefiore Medical Center
Locations (5):
- United States (5):
  - HealthAlliance Hospitals, Fitchburg, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albert Einstein Cancer Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York